CLINICAL TRIAL: NCT06346418
Title: Role of Maternal Effect Genes and Epimutations in Beckwith-Wiedemann Syndrome and Adverse Reproductive Outcomes
Brief Title: Maternal Genes and Epimutations: Beckwith-Wiedemann Syndrome & Reproductive Risks
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: Istituto Auxologico Italiano (Other); University of Campania Luigi Vanvitelli (Other); Federico II University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PNRR-MR1-2022-12376622
Record Dates: First submitted 2024-03-20; First posted 2024-04-04 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-01

CONDITIONS: Beckwith-Wiedemann Syndrome
MeSH Terms: conditions — Beckwith-Wiedemann Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- healthy women with offspring affected by BWS (Experimental): healthy women with offspring affected by BWS and peculiar reproductive history from our population of clinically and molecularly diagnosed BWS families
  Interventions: Genetic: WES analysis; Genetic: whole-genome methylation analysis
- women under 35 undergoing ART (Experimental): women under 35 undergoing ART for infertility (defined as failure to achieve a pregnancy after 12 months or more of regular unprotected sexual intercourses) and unable to obtain a live birth after three completed cycles or after the transfer of at least 6 blastocysts
  Interventions: Genetic: WES analysis; Genetic: whole-genome methylation analysis
- women under 35, with RPL (Experimental): women under 35, with RPL (defined as the loss of two or more pregnancies before 24 weeks of gestation)
  Interventions: Genetic: WES analysis; Genetic: whole-genome methylation analysis

INTERVENTIONS:
Genetic: WES analysis — Whole-exome sequencing will be performed as the first approach in all the recruited patients. First, we will analyze different subsets of genes, belonging to:
  1. Maternal effect genes as SCMC components and other related genes;
  2. Genes essential in the maturation of the oocyte and zygote progression through the early phases of the embryogenesis or highly expressed at different stages of oocyte maturation;
  3. Genes with known and potential roles in the establishment and control of genomic imprinting and involved in DNA methylation reactions.
  Subsequently, variants with a high pathogenicity score will be analyzed, to identify any genes that may be associated with the phenomenon, but do not belong to the previously described categories of genes. Finally, we will conduct a whole genome sequencing (WGS) analysis on a selected subgroup of BWS mothers with peculiar clinical histories and negative WES analysis, to explore all the noncoding and regulatory regions not targeted by WES.
Genetic: whole-genome methylation analysis — A whole-genome methylation analysis will be performed to identify methylation changes in women with reproductive problems including those with offspring affected by BWS

SUMMARY:
Pathogenic variants in subcortical maternal complex (SCMC) have been identified not only in mothers of Beckwith-Wiedemann syndrome (BWS) babies but also in women with reproductive disturbances such as failed pregnancy attempts and recurrent pregnancy loss. Based on the higher incidence of BWS in children born from Assisted Reproductive Technology (ART), this project aims to investigate incidence and molecular mechanism of pathogenic variants of SCMC in women with reproductive disorders. Study objectives will be (i) assess the incidence of these variants as a cause of differences in reproductive outcomes in the infertile female population and mothers of children with BWS; (ii) identify methylation changes in women with reproductive problems including those with offspring affected by BWS; (iii) determine the molecular causes underlying female infertility and imprinting disorder associated with damaging SCMC gene variants by employing a mouse model.

DETAILED DESCRIPTION:
The first aim of the project is to define the incidence of Maternal-Effect Genes (MEGs) and specifically of SCMC pathogenic variants as a cause of differences in reproductive outcomes in the infertile female population and mothers of BWS children. To this aim, three cohorts of patients will be recruited: healthy women with offspring affected by BWS and peculiar reproductive history from our population of clinically and molecularly diagnosed BWS families (Cohort 1), women under 35 undergoing ART for infertility (defined as failure to achieve a pregnancy after 12 months or more of regular unprotected sexual intercourses) and unable to obtain a live birth after three completed cycles or after the transfer of at least 6 blastocysts (Cohort 2), and women under 35, with RPL (Recurrent Pregnancy Loss defined as the loss of two or more pregnancies before 24 weeks of gestation) (Cohort 3).

To identify pathogenic variants, whole-exome sequencing (WES) will be performed as the first approach in all the recruited patients. WES analysis will be carried out following various steps. First, the investigators will analyze different subsets of genes, belonging to:

1. Maternal effect genes as SCMC components and other related genes;
2. Genes essential in the maturation of the oocyte and zygote progression through the early phases of the embryogenesis or highly expressed at different stages of oocyte maturation;
3. Genes with known and potential roles in the establishment and control of genomic imprinting and involved in DNA methylation reactions.

Subsequently, variants with a high pathogenicity score will be analyzed, to identify any genes that may be associated with the phenomenon, but do not belong to the previously described categories of genes. Finally, the investigators will conduct a whole genome sequencing (WGS) analysis on a selected subgroup of BWS mothers with peculiar clinical histories and negative WES analysis, to explore all the noncoding and regulatory regions not targeted by WES.

The second aim of this project is to employ whole-genome methylation analysis to identify methylation changes in women with reproductive problems including those with offspring affected by BWS. Specific tasks will be:

1. Determining the whole-genome methylation of blood leukocytes of the cohorts of women described in Aim 1 and comparing it with that of a similar number of sex- and age-matched controls;
2. Determining the whole-genome methylation of unfertilized oocytes derived from unsuccessful ART cycles of the same cohorts and comparing it with that of control oocytes (derived from either donation for research or public datasets).

DNA methylation will be determined in blood leukocytes by methylation array analysis and in unfertilized oocytes by single cell Bisulfite sequencing (scBS-Seq).

The third aim of the project is to determine the molecular mechanisms underlying female infertility and imprinting disorder associated with damaging SCMC gene variants by employing a mouse model. Specific tasks will be:

1. Determining the whole-genome methylation and RNA profiles of the Padi6 mut/mut oocytes and pre-implantation embryos obtained after IVF with wild-type sperm;
2. Transfer of the blastocysts derived from the IVF described in a) into pseudopregnant females and analysis of whole genome DNA methylation and RNA in the derived mid-gestation embryos by BS-seq and RNA-seq;
3. Mini-screening of epigenetics compounds on the 2-cell Padi6 mut/mut embryos. DNA methylation and RNA expression of the mouse oocytes and embryos will be determined by whole-genome scBS-seq and scRNA-seq.

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1: healthy women with offspring affected by BWS and peculiar reproductive history from our population of clinically and molecularly diagnosed BWS families;
* Cohort 2: women under 35 undergoing ART for infertility (defined as failure to achieve a pregnancy after 12 months or more of regular unprotected sexual intercourses) and unable to obtain a live birth after three completed cycles or after the transfer of at least 6 blastocysts;
* Cohort 3: women under 35, with RPL (defined as the loss of two or more pregnancies before 24 weeks of gestation).

Exclusion Criteria:

* presence of conventional and molecular karyotype alterations
* occurrence of known causes that can lead to decreased fertility or recurrent abortions: disorders of the ovaries, such as polycystic ovarian syndrome and other follicular disorders, disorders of the endocrine system causing imbalances of reproductive hormones levels, autoimmune conditions, male infertility, uterine or tubal dysfunctions and malformations, thrombophilic or noncorrected thyroid dysfunctions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
MEG Incidence | WES at specific genes in all the cohorts and SNP-array will be performed following enrollment and will be finalized within month 17. The last part related to WGS on a selected subgroup of BWS mothers will be accomplished from 16 to month 20
  Incidence of MEGs, particularly pathogenetic variants of SCMC, in infertile female population and mothers of children affected by BWS

SECONDARY OUTCOMES:
Compare DNA methylation | samples collected will be evaluated for whole-genome methylation within month 20
  Whole-genome DNA methylation of blood leukocytes of the cohorts of women with reproductive problems including those with offspring affected by BWS and comparing it with that of a similar number of sex- and age-matched controls. Bioinformatics analysis will be used to infer differentially methylated regions from methylation data and to classify women status based on methylation profiles. Due to the complex distribution associated with whole-genome methylation profiles, dimensionality reduction techniques (e.g. PCA,MDS) and clustering methods (both hierarchical and centroidbased) will be used to assess the importance of specific regions (e.g. imprinted loci) to discriminate prioritized women from controls according to their methylation profiles.
  with reproductive problems including those with offspring affected by BWS

CONTACTS AND LOCATIONS:
Overall Officials: Edgardo Somigliana, PhD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (2):
- Italy (2):
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Istituto Auxologico Italiano, Milan

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-20): https://cdn.clinicaltrials.gov/large-docs/18/NCT06346418/Prot_SAP_000.pdf